CLINICAL TRIAL: NCT06891261
Title: Evaluation of Endosseous Implants in One Stage Ridge Splitting Using the Conventional Technique Versus the Use of Piezo Surgery in the Maxilla
Brief Title: One Stage Ridge Splitting Using 2 Different Techniques in Maxilla
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mohannad Ahmed Ismail, Principle Investigator, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 00-0001-6142-0568
Record Dates: First submitted 2025-02-16; First posted 2025-03-24 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Ridge Augmentation; Bone Augmentation
Keywords: ridge augmentation; One stage ridge splitting in maxilla.; Piezo Surgery
MeSH Terms: interventions — Piezosurgery

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The patients were randomly allocated into two groups utilizing Random Allocation Software version 2.0. then the allocation was concealed in opaque sealed envelopes. In the study group (A) Piezo Surgery inserts are going to be used to create alveolar bone osteotomies, while in the control group (B) bone discs are used. All procedures were performed by one surgeon in both groups, the allocation was revealed to the operator just before the surgery. On the other hand, the patients, outcome assessor and the statistician who analyzed the collected data and performed the statistical analysis were blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study Group A: Piezo Surgery. (Active Comparator): Straight and angled bone inserts were utilized.
  Interventions: Device: Piezo Surgery.
- Control Group B: Conventional Technique. (Active Comparator): using bone discs of 7mm diameter mounted on contra angled 1:1 and 6.5mm diameter bone discs mounted on 1:1 external irrigation straight hand piece.
  Interventions: Procedure: Bone Discs.

INTERVENTIONS:
Device: Piezo Surgery. — Piezotome woodpecker®: Surgic touch.
  Arms: Study Group A: Piezo Surgery.
Procedure: Bone Discs. — bone discs mounted on staight hand piece and contra angled 1:1 gear ratio.
  Arms: Control Group B: Conventional Technique.

SUMMARY:
* The selected patients will be informed of the nature of the research work and informed consent will be obtained.
* Patients of both groups will be subjected to CBCT.
* Intra operative procedures (for both groups) followed by CBCT will be taken for every patient after 4 months.
* Infiltration local anesthesia will be given to the patient (Articaine 4% 1:100 000 epinephrine)

Both the study and control group will receive:

* In Recipient site, full thickness mucoperiosteal flap pyramidal flap, reflection using mucoperiosteal elevator.
* The defective site is reevaluated.
* Flap advancement inorder to allow tension free flap closure.
* In the Study group: Piezo surgery bone inserts is used to cut crestal osteotomies.
* In the Control group: Bone discs diameter is used.
* Followed by, the use of bone chisels.
* The point and pilot implant drills are used followed by bone expanders. Based on the preexisting bone, the defect morphology and bone quality. The implant is submerged below the alveolar crest to compensate for crestal bone resorption.
* Following partial immobilization of the buccal bone segment either book or island pattern. The fixture is inserted submerged below the alveolar bone crest.

Followed by bone smoothening and roundation under external saline irrigation at recommended speed of 38000rpm and gear ratio 1:1 calibrated on fesiodespenser.

* Xenogenic bone particle size of 0.5 mm to 1mm is going to be condensed into the dead space.
* Recheck adequate flap advancement to allow tension free closure.
* Double line closure using horizontal mattress followed by interrupted sutures to allow contact area and wound edge eversion.

DETAILED DESCRIPTION:
* The selected patients will be informed of the nature of the research work and informed consent will be obtained then randomized in equal proportions between control group conventional ridge splitting and study ridge splitting using piezo surgery.
* Patients of both groups will be subjected to CBCT (diagnostic for upper arch), diagnostic wax-up and stent fabrication.
* Intra operative procedures (for both groups) followed by CBCT will be taken for every patient after 4 months.
* Scrubbing and draping of the patient will be carried out in a standard fashion for intra oral procedures.
* Infiltration local anesthesia will be given to the patient (Articaine 4% 1:100 000 epinephrine)

Both the study and control group will receive:

* In Recipient site, using 15C blade on Bard Parker handle incision of full thickness mucoperiosteal flap inorder to obtain, three-line pyramidal flap, reflection using mucoperiosteal elevator molt 9.
* The defective site is reevaluated after its primary evaluation on CBCT using UNC periodontal probe.
* Flap advancement using periosteal releasing incision inorder to allow later tension free flap closure.
* In the Study group: Piezo surgery bone inserts is used to cut crestal osteotomy in the center of the alveolar bone ridge bucco-lingual traversing the compact bone into the spongiosa Followed by two semi vertical osteotomies at least 1.5mm away from the adjacent teeth.
* In the Control group: Bone discs diameter 7mm mounted on contra angled 1:1 is used to cut crestal osteotomy in the center of the alveolar bone ridge bucco-lingual traversing the compact bone into the spongiosa Followed by two semi vertical osteotomies at least 1.5mm away from the adjacent teeth using bone discs diameter 6.5mm mounted on external irrigation straight hand piece.
* First, the spatula bone chisels are used to make sure of extension of osteotomies into the spongy bone in addition to, adequate free of the cut corners, followed by sequential use of tapered bi-angled bone chisels and hammering with bone mallet 3mm shorter than the length of the proposed implant to gain adequate 1ry stability with concurrent support of the buccal plate of bone.
* The point and pilot implant drills are used followed by the sequential use of bone expanders diameters 2.6, 3, 3.4, 3.8 to place an implant of diameter 3.7 or 4.1mm. Based on the preexisting bone, the defect morphology and bone quality. The implant is submerged about 2mm to 3mm below the alveolar crest to compensate for crestal bone resorption.
* Following partial immobilization of the buccal bone segment either book or island pattern. The fixture is inserted submerged below the alveolar bone crest by 2mm to 3mm. Followed by bone smoothening and roundation using large round diamond stone mounted on straight hand piece with external saline irrigation at recommended speed of 38000rpm and gear ratio 1:1 calibrated on fesiodespenser. To avoid soft tissue irritation.
* Xenogenic bone particle size of 0.5 mm to 1mm is going to be condensed into the dead space. To act as a scaffold for the formation of autogenous bone.
* Recheck adequate flap advancement by visualizing passive flap approximation, to allow tension free closure.
* Double line closure using horizontal mattress placed 5mm away from flap margins followed by interrupted sutures on top to allow contact area which is preferred to point contact and wound edge eversion.

ELIGIBILITY:
Inclusion Criteria:

* Patients with maxilla residual alveolar bone height not less than 8 mm.
* Alveolar bone width from 5mm to 3mm.
* Both genders.
* At least single missing tooth.
* Previous failed implants.
* Tapered or cylinder cross sectioned alveolar bone defect pattern.

Exclusion Criteria:

* Heavy smokers more than 20 cigarettes per day.
* Patients with bone disease that may affect normal healing, example; hyperparathyroidism.
* Patients had radiotherapy and chemotherapy in head and neck.
* Patients had neoplasms in sites to be grafted.
* Patients with Metabolic diseases uncontrolled diabetic patients, Glycated hemoglobin (Hb A1c) more than 7 mg\dl.
* Pregnant females.
* Patients with Para functional habits, apprehensive and non-cooperative.
* Bone pathology related to the site to be grafted.
* Psychological problems, stress situation (socially or professionally), emotional instability, and unrealistic patients' expectations.
* Intraoral soft and hard tissue pathology.
* Systemic condition that contraindicates implant placement.
* Under the age of 18 years.
* Hourglass defects or defects with bone concavities and or undercuts.

Ages: 20 Years to 48 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2025-07-30 (Estimated); Study Completion 2025-10-31 (Estimated)

PRIMARY OUTCOMES:
Bone Quality of bone gain. | At 4 months from ridge augmentation.
  Measured using linear measurements from CBCT in millimeters.

SECONDARY OUTCOMES:
Soft Tissue Dehiscence. | Baseline 1st Week.
  Exposure of the augmented site. Written Binary Numerical.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Spin-Neto R, Landazuri Del Barrio RA, Pereira LA, Marcantonio RA, Marcantonio E, Marcantonio E Jr. Clinical similarities and histological diversity comparing fresh frozen onlay bone blocks allografts and autografts in human maxillary reconstruction. Clin Implant Dent Relat Res. 2013 Aug;15(4):490-7. doi: 10.1111/j.1708-8208.2011.00382.x. Epub 2011 Aug 11. PMID 21834864
- [Background] Acocella A, Bertolai R, Ellis E 3rd, Nissan J, Sacco R. Maxillary alveolar ridge reconstruction with monocortical fresh-frozen bone blocks: a clinical, histological and histomorphometric study. J Craniomaxillofac Surg. 2012 Sep;40(6):525-33. doi: 10.1016/j.jcms.2011.09.004. Epub 2011 Nov 9. PMID 22075326
- [Background] Dasmah A, Thor A, Ekestubbe A, Sennerby L, Rasmusson L. Particulate vs. block bone grafts: three-dimensional changes in graft volume after reconstruction of the atrophic maxilla, a 2-year radiographic follow-up. J Craniomaxillofac Surg. 2012 Dec;40(8):654-9. doi: 10.1016/j.jcms.2011.10.032. Epub 2011 Dec 3. PMID 22137760
- [Background] AlGhamdi AS. Post-surgical complications of symphyseal block graft with and without soft tissue grafting. Saudi Med J. 2013 Jun;34(6):609-15. PMID 23756926
- [Background] Monje A, Monje F, Chan HL, Suarez F, Villanueva-Alcojol L, Garcia-Nogales A, Wang HL. Comparison of microstructures between block grafts from the mandibular ramus and calvarium for horizontal bone augmentation of the maxilla: a case series study. Int J Periodontics Restorative Dent. 2013 Nov-Dec;33(6):e153-61. doi: 10.11607/prd.1664. PMID 24116370
- [Background] Aloy-Prosper A, Penarrocha-Oltra D, Penarrocha-Diago M, Penarrocha-Diago M. The outcome of intraoral onlay block bone grafts on alveolar ridge augmentations: a systematic review. Med Oral Patol Oral Cir Bucal. 2015 Mar 1;20(2):e251-8. doi: 10.4317/medoral.20194. PMID 25662543
- [Background] Reininger D, Cobo-Vazquez C, Monteserin-Matesanz M, Lopez-Quiles J. Complications in the use of the mandibular body, ramus and symphysis as donor sites in bone graft surgery. A systematic review. Med Oral Patol Oral Cir Bucal. 2016 Mar 1;21(2):e241-9. doi: 10.4317/medoral.20938. PMID 26827063
- [Background] Khoury F: Augmentation of severe bony defects with intraoral bone grafts: biological approach and long-term results J Oral Maxillo Fac Surg 2017Volume 46, Supplement 1, Pages 26-27.
- [Background] Claudino M, Julio C L, Luis E M, Bernardo M, Fernando G, tomographic evaluation of atrophic maxilla rehabilitated with autogenous and xenogeneic block grafts. Journal of Research in Dentistry 2017, 4(4):112-117.